CLINICAL TRIAL: NCT00978913
Title: Evaluation of Dendritic Cells Transfected With Survivin, hTERT and p53 mRNA as a Treatment for Patients With Metastatic Breast Cancer or Malignant Melanoma
Brief Title: Transfected Dendritic Cell Based Therapy for Patients With Breast Cancer or Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA 0914
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer; Malignant Melanoma
Keywords: dendritic cell; cancervaccine; breast cancer; malignant melanoma; Cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms; Melanoma | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC vaccination and Cyclophosphamide (Experimental)
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — DC vaccination, one vaccine biweekly
  Other Names: dendritic cell vaccine; Cyclophosphamide, Sendoxan®, Baxter

SUMMARY:
The primary aim of this study is to evaluate the toxicity of the vaccine and the combination of the vaccine and Cyclophosphamide, and to evaluate the immune response induced by the vaccine. The secondary aim is to investigate the clinical tumour response and duration of tumour and immune response.

DETAILED DESCRIPTION:
Phase I trial. Single center study; patients will be referred to the study center from other institutions in Denmark. 14 patients will be included in this phase I trial DC vaccination regime consists of primary 6 biweekly intradermal injections with transfected dendritic cells, followed by monthly injections until progression; Cyclophosphamide is used as vaccine adjuvant.

Defined procedures are employed for generation of autologous dendritic cells for clinical application in a classified laboratory. Unmobilized leukapheresis will be used for isolation of large-scale mononuclear cells, and dendritic cells will be generated from monocytes by cytokine stimulation and transfected with mRNA encoding for hTERT, survivin and p53 if the tumour express p53. Frozen preparations of dendritic cells will be prepared using automated cryopreservation. Each patient will receive a minimum of 1x106 dendritic cells per treatment supplemented with Cyclophosphamide 50 mg twice a day every second week. Toxicity including autoimmunity will be evaluated using the Common Toxicity Criteria (CTC).

ELIGIBILITY:
Inclusion Criteria:

1. Histological verified metastatic breast cancer or malignant melanoma, in progression
2. ≥ 18 years
3. the patient must be habil
4. Performance status ≤ 1 on Zubrod-ECOG-WHO-scale
5. Leukocytes and platelets must be ≥normal. Hg ≥ 6.0
6. creatinin must be normal
7. Liverparametre <2.5 x normal. Bilirubin <30
8. Expected survival > 3 months
9. Informed consent

11. At least one measurable lesion according to RECIST criteria.

Exclusion Criteria:

1. Indication for chemotherapy
2. Other malignancies
3. Brain metastases
4. severe medical condition
5. Acute/chronic infection with ex. HIV, hepatitis, tuberculose
6. Severe allergy
7. Autoimmune disease
8. Other treatment with immune suppressing agents, other anticancer agents or experimental drugs
9. Uncontrolled hypercalcemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
to evaluate the toxicity of the vaccine in combination with Cyclophosphamide | biweekly

SECONDARY OUTCOMES:
to investigate the clinical tumor response and the duration | after 12 weeks
to evaluate the duration of tumor and immunoresponse | 3, 6, 9 months
to evaluate immune response | at 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, prof.MD, Study Director — Department of Oncology, Herlev University Hospital, Herlev Ringvej 75,2730 Herlev
Locations (1):
- Department of Oncology, Herlev University Hospital, Herlev, Denmark